CLINICAL TRIAL: NCT05111119
Title: Making PrEP Smart: An HIV Testing and PrEP Electronic Support Tool ("SmartPrEP" App) for Women on PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAT7092
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: HIV/AIDS
Keywords: Pre-Exposure Prophylaxis (PrEP); HIV Prevention; Mobile App
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Making PrEP Smart (Experimental): The Making PrEP Smart intervention is a mobile-based application which provides PrEP adherence reminders and supports HIV-self and partner testing for cis- and transgender women.
  Interventions: Behavioral: Making PrEP Smart

INTERVENTIONS:
Behavioral: Making PrEP Smart — The Making PrEP Smart intervention is a mobile-based application with the following components:
  * Notification-based PrEP Reminders and Adherence Self-Monitoring
  * HIV self-testing facilitation, interpretation of results, and testing support
  * HIV partner testing facilitation, interpretation of results, and testing support
  * Nearby HIV clinic contact information

SUMMARY:
Primary Objective: To assess PrEP adherence among sexually-active and/or injection-drug using, HIV-negative cis- and transgender women who use the "SmartPrEP" phone app to support PrEP adherence during a 12-month period of observation.

Secondary Objective: To assess the acceptability of using the SmartPrEP app to support HIV self-testing and partner testing among sexually active and/or injection-drug using, HIV-negative cisgender and transgender women on PrEP.

Exploratory Objectives: To describe patterns of PrEP adherence and user feedback on acceptability, utility, and features of the app; To assess correlations between self-reported sexual behavior and PrEP adherence; To assess patterns of HIV testing (self and partner testing), self-reported reasons for HIV testing, and correlations with test results.

DETAILED DESCRIPTION:
The purpose of this study is to understand if a smartphone app, SmartPrEP, will help promote HIV self-testing and PrEP adherence among cisgender and transgender women over a twelve-month period. As part of this, participants will be required to download the SmartPrEP app and participate in six study visits starting at enrollment, Month 1, Month 3, Month 6, Month 9, and Month 12. Most visits will take place at the Bronx Prevention Center and include adherence counseling, app acceptability assessments, behavioral risk assessments, and STI/HIV testing. App data will be collected which evaluates PrEP adherence, HIV self-testing, and HIV partner testing. Additionally, all participants will be invited to take part in either a focus group discussion (FGD) or an open-ended, in-depth interview (IDI) to elicit their thoughts and preferences regarding the SmartPrEP app acceptability. Interventions consist of (1) smartphone app "SmartPrEP"; (2) PrEP medication.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older (confirmed by ID)
* self-identify as either a cisgender or transgender woman
* eligible for and willing to initiate PrEP or already on PrEP [having initiated PrEP within the last three months per participant self-report]
* documented negative HIV test result at Screening Visit
* Has a mobile phone with a minimum of 3G network with an active cellular plan
* no signs/symptoms of acute HIV infection
* normal renal function (eCrCl of >/= 60 ml/min)
* not taking contraindicated medications
* documented negative hepatitis B virus (HBVAg) status or documented evidence of seroimmunity
* if HCV Ab positive, documented evidence of previous completed treatment, resolution of active HCV infection (i.e. documented negative HCV RNA), or documented evidence of PCP/HCV care provider management/treatment progress
* meets CDC criteria for HIV risk
* willing to complete all required study procedures including the use of Truvada.

Exclusion Criteria:

* age under 18 years;
* HIV-positive status based on documented test results at at Screening or Enrollment Visits;
* any sign or symptom of acute HIV infection at screening or enrollment visit, until HIV status is confirmed negative via HIV RNA PCR testing;
* renal function, eCrCl< 60 mL/min at Screening or Enrollment visit;
* inability to provide informed consent;
* pregnancy or breast-feeding;
* plans to move away from NYC area in the next 12-month period;
* Current use of HIV post-exposure prophylaxis (PEP), though participants who wish to transition from PEP to PrEP will be eligible at the completion of PEP
* Continued need for/use of medications with potential for adverse interactions with Truvada (FTC/TDF) or Descovy (TAF/FTC) on a case-by-case basis, i.e., hepatitis C antiviral agents, such as EPCLUSA (sofosbuvir/velpatasvir) or VOSEVI (sofosbuvir/velpatasvir/voxilaprevir); NRTIs, such as didanosine; medications that may decrease renal function (i.e., high-dose or multiple NSAIDS, aminoglycosides; and other medications that may result in compromising a participant's overall health if combined with Truvada, per the discretion of the IOR;
* History of self-reported low adherence to PrEP, based on study team's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on self-representation of gender identity. Participants must identify as a cis- or transgender woman.
Enrollment: 53 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with optimal PrEP adherence | 12-month period of observation
  This is to measure PrEP Adherence, defined as taking >/= 6 doses per week, as recorded in the SmartPrEP app.

SECONDARY OUTCOMES:
Proportion of participants who perform HIV self-testing | 12-month period of observation
  This is to measure HIV Self-Testing, as recorded in the SmartPrEP App during the study. Participant-reported reasons for performing HIV self-testing will be included in the analyses.
Proportion of participants who rated app to be acceptable | 12-month period of observation
  This is to measure acceptability of the SmartPrEP App, per participant report, as collected in the focus group discussions and in-depth interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Justman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States